CLINICAL TRIAL: NCT03286309
Title: Soft Robotic Hand System for Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.396-T
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG-driven soft robot hand (Experimental): subjects will receive EMG-driven soft robot hand system.
  Interventions: Device: soft robot hand system
- sham group (Placebo Comparator): subjects will receive passive pre-programmed soft robot hand system.
  Interventions: Device: soft robot hand system

INTERVENTIONS:
Device: soft robot hand system — subjects will wear the soft robot hand system and receive 60 minutes (including preparation time) hand exercise.

SUMMARY:
The soft robotic system could provide objective and quantifiable measures of subject performance. By combining voluntary motor intention and the robotic hand technology, the system will facilitate the recovery process of stroke patients.

ELIGIBILITY:
Inclusion criteria:

1. at chronic stage (6 months after the onset of stroke) with a pure unilateral motor paresis after a stroke (ischemic or hemorrhagic);
2. sufficient cognition to follow simple instructions as well as understand the content and purpose of the study;
3. able to sit up for 45 minutes (with or without assistance).

Exclusion criteria:

1. Patients with severe dysphasia (either expressive or comprehensive) with inadequate communication;
2. any additional medical or psychological condition affecting their ability to comply with the study protocol;
3. history of other neurological disease, psychiatric disorder, including alcoholism and substance abuse.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Upper limb Fugl Meyer Assessment | 3-month follow up

SECONDARY OUTCOMES:
Action Research Arm Test | 3-month follow up
Modified Ashworth Scale | 3-month follow up
  Scale from 0 to 4, whereas 0 is no increase in tone and 4 is limb rigid in flexion or extension
Box and Block Test | 3-month follow up
Max Voluntary Grip Force | 3-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi XQ, Ti CE, Lu HY, Hu CP, Xie DS, Yuan K, Heung HL, Leung TW, Li Z, Tong RK. Task-Oriented Training by a Personalized Electromyography-Driven Soft Robotic Hand in Chronic Stroke: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2024 Aug;38(8):595-606. doi: 10.1177/15459683241257519. Epub 2024 May 29. PMID 38812378